CLINICAL TRIAL: NCT07375394
Title: Evaluation of a 3D-Printed Extraoral Camera Assembly for Standardization of Dental Photography: Randomized Controlled Clinical Trial
Brief Title: 3D-Printed Extraoral Camera for Standardized Dental Photography
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer, Department of Periodontology, Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: 12.2025
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Malnutrition
Keywords: undergraduate medical students; dental nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates whether a 3D-printed extraoral camera assembly can improve the reproducibility and dimensional consistency of dental photographs compared with conventional DSLR methods. By standardizing camera position, distance, and angle, the assembly provides a non-contact, operator-independent approach to ensure consistent image geometry, supporting more accurate clinical records, esthetic documentation, and digital analyses.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate dental students
* Egyptian nationality
* Both genders

Exclusion Criteria:

* Postgraduate dental students
* Incomplete questionnaires
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include undergraduate dental students of Egyptian nationality, encompassing both genders. Excluded from participation are postgraduate dental students, individuals who submit incomplete questionnaires, and those who decline to participate.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
knowledge | 3 months
  Knowledge score regarding dental nutrition

SECONDARY OUTCOMES:
Attitude score | 3 months